CLINICAL TRIAL: NCT00537940
Title: A Randomized, Double-blind, Parallel-group Multi-center Comparative Flexible-dose Trial Of Pregabalin Versus Gabapentin As Adjunctive Therapy In Subjects With Partial Seizures.
Brief Title: Comparative Study Of Pregabalin And Gabapentin As Adjunctive Therapy In Subjects With Partial Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081143; 2007-003161-40 (EudraCT Number); 207103 (Other: Alias Study Number)
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-11

CONDITIONS: Epilepsy; Partial Seizure Disorder; Epilepsies, Partial; Complex Partial Seizure Disorder
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Epilepsy, Complex Partial | interventions — Pregabalin; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Pregabalin
- B (Active Comparator)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Pregabalin — 150, 300, 450 mg/day administered orally TID, until seizure control/improvement or intolerable side effects
  Arms: A
Drug: Gabapentin — 300, 600, 1200, 2000 mg/day administered orally TID, until seizure control/improvement or intolerable side effects
  Arms: B

SUMMARY:
To compare the efficacy of pregabalin and gabapentin, as adjunctive therapy in subjects with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) must be > 18 years or ≤ 80 years of age, with a diagnosis of epilepsy with partial seizures, as defined in the International League Against Epilepsy (ILAE) classification of seizures; partial seizures may be simple or complex, with or without secondary tonic-clonic generalization.
* Subjects must be have been diagnosed with epilepsy for at least 2 years, and must have been unresponsive to treatment with at least two but no more than five prior antiepileptic drugs (AEDs), and at the time of study enrollment are on stable dosages of 1 or 2 standard AEDs.
* They must have had a 12 lead electrocardiogram (ECG) without clinically significant abnormal findings prior to randomization.
* Subjects must have had magnetic resonance imaging or contrast enhance computed tomography scan of the brain that demonstrated no progressive structural central nervous system abnormality at the time of the diagnosis of epilepsy.
* Women of childbearing potential must be established on an effective method of contraception during the study. Women should also have a negative pregnancy test prior to study entry.
* During the 6-week baseline period, subjects must have had a minimum of four partial seizures, with no 28 day period free of partial seizures with or without secondary generalization. A caregiver or witness must be with the subject for a sufficient duration to accurately chronicle the occurrence of seizures. These seizures must have been documented in the subject's diary.
* Subjects with electroencephalograph (EEG) testing done within 2 years of randomization. EEG abnormalities should be consistent with a diagnosis of focal-onset epilepsy.
* Signed and dated informed consent will be obtained from each subject (only include those able to consent) in accordance with the local regulatory and legal requirements.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures. Subjects who are willing, but need assistance for self administered questionnaires may be considered acceptable, but must first be discussed on a case-by-case basis with the Pfizer monitor prior to any to any screening tests or procedures for the study.

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or intending to become pregnant during the course of the trial.
* Subjects with other neurologic illness that could impair endpoint assessment, or patients with Lennox-Gastaut syndrome, absence seizures, status epilepticus within the 12 months prior to study entry, or with seizures due to an underlying medical illness or metabolic syndrome.
* Subjects with clinically significant liver disease or with a calculated creatinine clearance of <60mL/min.
* Subjects with a history of lack of response, hypersensitivity or poor tolerability to gabapentin or pregabalin.
* Previous use of gabapentin or pregabalin within 2 weeks prior to screening or likelihood of engaging in these treatments during the study period.
* Use of prohibited medications as listed in the protocol in the absence of appropriate washout phase or the likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.
* Participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
* Subjects who are not suitable to be treated with pregabalin or gabapentin according to the respective local labeling.
* Subjects with a history of retinal abnormalities or treatment with retinotoxic agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2008-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Hospital Clinica Biblica, San José, Costa Rica
- El Salvador (2):
  - Instituto de Neurociencias, San Salvador
  - Clinica de Especialidades Neurologicas, San Salvador
- Guatemala (2):
  - Private Office, Guatemala Ciudad, Departamento de Guatemala
  - Private Office, Guatemala City
- Peru (3):
  - Clinica Anglo Americana, Lima
  - Torre de Consultorios Clinica Anglo Americana, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen - Essalud, Lima

REFERENCES:
- [Derived] French J, Glue P, Friedman D, Almas M, Yardi N, Knapp L, Pitman V, Posner HB. Adjunctive pregabalin vs gabapentin for focal seizures: Interpretation of comparative outcomes. Neurology. 2016 Sep 20;87(12):1242-9. doi: 10.1212/WNL.0000000000003118. Epub 2016 Aug 12. PMID 27521437
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081143&StudyName=Comparative%20Study%20Of%20Pregabalin%20And%20Gabapentin%20As%20Adjunctive%20Therapy%20In%20Subjects%20With%20%20Partial%20Seizures

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 561 participants were screened and 482 participants participated in the study; 242 participants were randomized but one participant from the pregabalin group and one participant from the gabapentin group were not treated. Hence 241 participants were treated in each treatment group. Participants were randomized at 56 centers.
Pre-assignment Details: One participant from the pregabalin group and one participant from the gabapentin group were randomized but not treated.
Groups:
- Pregabalin: Pregabalin was initiated at 150 mg/day [50 mg capsules orally three times a day (TID)] for 1 Week followed by pregabalin 300 mg/day (100 mg TID) orally TID up to Week 5 in the Titration Phase (TP). Participants who had adequate seizure control (adequate: >=50% reduction in seizures) with acceptable tolerability with pregabalin 300 mg/day in TP, continued same dose until the end of TP (Week 9) and then entered the maintenance phase (MP) on this dose. If seizure control was inadequate, the pregabalin dose was escalated to 450 mg/day orally (150 mg TID) from Weeks 5 through 9. If the participants had adequate seizure control with acceptable tolerability on this dose, then they entered the MP on this dose. If there was inadequate seizure control at the end of Week 9, the dose was escalated a final time to 600 mg/day (200 mg TID) at which time they entered the MP.
- Gabapentin: Gabapentin was initiated at 300 mg/day [100 mg capsules orally three times a day (TID)] followed by gabapentin 600 mg/day (200 mg TID) on Day 3. At the end of Week 1 (Day 7), the dose was increased to 1200 mg/day (400 mg TID) and remained on this dose for the next 4 weeks). Participants who had adequate seizure control (>=50% reduction in seizure frequency) with acceptable tolerability during this initial 5-week period, remained on this dose until the end of theTP (Week 9), then entered the MP on this dose. If seizure control was inadequate, the gabapentin dose was escalated to 1500 mg/day (500 mg TID) during Weeks 5 through 9. If they had adequate seizure control with acceptable tolerability on this dose, they entered the MP on this dose. If there was inadequate seizure control at the end of Week 9, the dose was escalated a final time to 1800 mg/day (600 mg TID), at which time they entered the MP.
Period: Overall Study
Arm/Group | Pregabalin | Gabapentin
Started | 241 | 241
Completed Titration Phase | 213 | 210
Completed Maintenance Phase | 187 | 172
Entered Opt Blinded Continuation Phase | 140 | 139
Completed | 58 (2 participants had both treatment related and non-treatment related AE leading to discontinuation.) | 62
Not Completed | 183 | 179
Not completed — Adverse Event | 20 | 19
Not completed — Lack of Efficacy | 8 | 16
Not completed — Lost to Follow-up | 23 | 29
Not completed — Withdrawal by Subject | 113 | 95
Not completed — Protocol Violation | 6 | 4
Not completed — Pregnancy | 1 | 1
Not completed — Study terminated by sponsor | 2 | 3
Not completed — Other | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Gabapentin | Total
Number analyzed (Participants) | 241 | 241 | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (13.0) | 35.3 (12.9) | 35.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 111 | 225
  Male | 127 | 130 | 257

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 28-day Seizure Frequency at Week 21.
Description: The seizures were recorded by the participants, by a family member, by a caregiver, or by a legal guardian and documented in a daily seizure diary. Participant's 28-day seizure frequency of all partial seizure was assessed during double blind (TP + MP) phase compared with baseline. Total partial seizure is defined as the total number of (simple partial seizure + complex partial seizure + secondary generalized tonic clonic seizure [SGTC]).
Time Frame: 6 weeks Baseline, 21 weeks through End of MP for 27 weeks
Population: Full analysis set (FAS) included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation.
Measure: Median (Full Range); unit: percent change
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 238 | 240
percent change | -58.65 [-100.0 to 180.0] | -57.43 [-100.0 to 392.4]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Rank analysis of covariance (ANCOVA) model was used to derive p-value with treatment as main effect and cluster as cofactor, percent change in 28-day seizure counts between Baseline and treatment periods as dependent variable. Median differences and 95% confidence interval (CI) were based on Hodges-Lehmann estimation; Test type: Superiority or Other; p = 0.8708, Ranked ANCOVA; Median Difference (Final Values) = 0.0, 95% CI 2-sided [-6.0 to 7.0]

2. Secondary Outcome: Percentage of Participants With 50% Reduction From Baseline in 28-day Seizure Rate at Week 21.
Description: Participants who had at least 50% reduction in seizure frequency from Baseline to double-blind treatment (TP + MP) were considered as 50% responders. If percent change from baseline <= -50 then responder rate = 1 (yes) otherwise responder rate = 0 (no).
Time Frame: 6 weeks Baseline, 21 weeks through End of MP for 27 weeks
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 Baseline and post Baseline primary efficacy evaluation. n=is the number of subjects that can be analyzed for each treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 238 | 240
Percentage of participants
  All Partial Seizure (n=238, 240) | 56.3 [50.0 to 62.6] | 58.3 [52.1 to 64.6]
  Simple Partial (n=87, 88) | 55.2 [44.7 to 65.6] | 53.4 [43.0 to 63.8]
  Complex Partial (n=161, 158) | 56.5 [48.9 to 64.2] | 55.1 [47.3 to 62.8]
  SGTC (n=112, 114) | 50.9 [41.6 to 60.2] | 60.5 [51.6 to 69.5]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; The odds ratio and its 95% CI are calculated by exponentiating the log odds ratio and 95% CI that correspond to the treatment contrast in the logistic regression model with treatment as fixed effect and Baseline term and country as covariate. All statistical tests for secondary efficacy parameters were two sided and performed at significance level of α = 0.05. The above statistical analysis applies to All Partial Seizures - FAS Population; Test type: Superiority or Other; p = 0.662, Regression, Logistic; Odds Ratio (OR) = 0.920, 95% CI 2-sided [0.635 to 1.335]

3. Secondary Outcome: Percentage of Participants With 75% Reduction From Baseline in 28-day Seizure Rate at Week 21.
Description: Participants who had at least 75% reduction in seizure frequency from Baseline to double-blind treatment (TP + MP) were considered as 75% responders. If percent change from baseline <= -75 then 75% responder rate = 1 (yes) otherwise responder rate = 0 (no). Total partial seizure is defined as the total number of (simple partial seizure + complex partial seizure + SGTC).
Time Frame: 6 weeks Baseline, 21 weeks through End of MP for 27 weeks
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 Baseline and post Baseline primary efficacy evaluation. n=is the number of participants that can be analyzed for each treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 238 | 240
Percentage of participants
  All Partial Seizure (n=238, 240) | 33.6 [27.6 to 39.6] | 34.2 [28.2 to 40.2]
  Simple Partial (n=87, 88) | 36.8 [26.7 to 46.9] | 33.0 [23.1 to 42.8]
  Complex Partial (n=161, 158) | 37.3 [29.8 to 44.7] | 36.1 [28.6 to 43.6]
  SGTC (n=112, 114) | 38.4 [29.4 to 47.4] | 43.9 [34.8 to 53.0]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.9232, Fisher Exact — All partial seizure: p-value was calculated from the 2-sided Fisher's exact test
Statistical Analysis 2: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.6361, Fisher Exact — Simple Partial: p-value was calculated from the 2-sided Fisher's exact test
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.9075, Fisher Exact — Complex partial: p-value was calculated from the 2-sided Fisher's exact test
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.4203, Fisher Exact — SGTC seizure: p-value was calculated from the 2-sided Fisher's exact test

4. Secondary Outcome: Percentage of Participants Without Seizures.
Description: Seizure free for 28 days was defined as participants who have not experienced any seizure (simple partial, complex partial and SGTC) for at least 28 consecutive days from their last seizure until the end of the MP. Same participant could be seizure free for a specific type of seizure but not necessarily for the other types of seizure.
Time Frame: 6 weeks Baseline, 21 weeks through End of MP for 27 weeks
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 Baseline and post Baseline primary efficacy evaluation. N (number of participants analyzed)=participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 189 | 182
percentage of participants
  All Partial Seizure (n=189, 182) | 30.7 [24.1 to 37.3] | 34.1 [27.2 to 41.0]
  Simple Partial (n=74, 66) | 29.7 [19.3 to 40.1] | 36.4 [24.8 to 48.0]
  Complex Partial (n=126, 123) | 37.3 [28.9 to 45.8] | 40.7 [32.0 to 49.3]
  SGTC (n=95, 91) | 46.3 [36.3 to 56.3] | 42.9 [32.7 to 53.0]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.5069, Fisher Exact — All partial seizure: p-value was calculated from the 2-sided Fisher's exact test
Statistical Analysis 2: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.4721, Fisher Exact — Simple partial seizure: p-value was calculated from the 2-sided Fisher's exact test
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.6054, Fisher Exact — Complex partial seizure: p-value was calculated from the 2-sided Fisher's exact test
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.6603, Fisher Exact — SGTC seizure: p-value was calculated from the 2-sided Fisher's exact test

5. Secondary Outcome: Change From Baseline in the 28-day Secondarily Generalized Tonic-clonic (SGTC) Seizure Frequency at Week 21.
Description: Change in SGTC = (Proportion of SGTC/All Partial Seizure rate during at the double-blind phase) - (Proportion of SGTC/All Partial Seizure rate at Baseline). Negative values indicate reduction from baseline.
Time Frame: 6 weeks Baseline, 21 weeks through End of MP for 27 weeks
Population: SGTC population included all participants who had at least 1 SGTC seizure during either Baseline or double-blind phase. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: percentage of all partial seizure/28days
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 114 | 114
percentage of all partial seizure/28days
  Baseline (n=114, 114) | 56.53 (40.856) | 59.60 (40.571)
  Change from Baseline at Double Blind (n=104, 98) | 1.59 (28.164) | -2.17 (26.024)

6. Secondary Outcome: Reduction in Proportion of the 28-day SGTC Seizure Rate Over the Total Partial Seizure Rate at Week 21.
Description: SGTC Responder is defined as a participant who shows reduction from Baseline to double-blind phase in proportion of 28-Day SGTC Seizure Rate to 28-Day All Partial Seizure Rate.
Time Frame: 6 weeks Baseline, 21 weeks through End of MP for 27 weeks
Population: SGTC population included all participants who had at least 1 SGTC seizure during either Baseline or double-blind phase. n is the number of participants analyzed for SGTC. Twenty-six participants were not included in the n because they did not have a post Baseline all partial seizure, but they were included in the analysis by seizure type.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 104 | 98
percentage of responders | 30.8 [21.9 to 39.6] | 39.8 [30.1 to 49.5]
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Test type: Superiority or Other; p = 0.1881, Fisher Exact — p-value is calculated using Fisher Exact Test

7. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Score.
Description: HADS: participant rated questionnaire with 2 subscales. Hospital Anxiety and Depression Scale - anxiety (HADS-A) assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); Hospital Anxiety and Depression Scale - depression (HADS-D) assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 21
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation. N (number of participants analyzed)=participants who were evaluable for this measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 238 | 240
Units on a scale
  Baseline HADS-A (n=238, 240) | 7.82 (0.31) | 7.60 (0.31)
  HADS- A Change at Week 21/ET (n=212, 210) | -0.92 (0.26) | -0.83 (0.27)
  Baseline HADS-D (n=238, 240) | 5.94 (0.29) | 5.65 (0.29)
  HADS-D Change at Week 21/ET (n=212, 210) | -0.59 (0.24) | -0.42 (0.24)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Baseline, HADS-A: ANCOVA model was used to calculate least square (LS) mean estimates of the treatment difference along with 95% CI, with main effects of treatment and and country as covariates; Test type: Superiority or Other; p = 0.5643, ANCOVA; LS Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.53 to 0.97], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Pregabalin vs Gabapentin; Change at Week 21 / ET , HADS-A: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country as covariates; Test type: Superiority or Other; p = 0.7712, ANCOVA; LS Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.73 to 0.54], Standard Error of Mean 0.32
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin; Baseline, HADS-D: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.4236, Ranked ANCOVA; LS Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.41 to 0.97], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin; Change at Week 21/ET, HADS-D: ANCOVA model was used to calculate LS mean estimates of the treatment1difference along with 95% CI, with main effects of treatment and combined center, and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.5492, Ranked ANCOVA; LS Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.75 to 0.40], Standard Error of Mean 0.29

8. Secondary Outcome: Medical Outcomes Study Sleep Scale (MOS-SS) Score.
Description: Participant-rated 12-item questionnaire to assess constructs of sleep over past week; 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence (range:0-100); sleep quantity (range:0-24), optimal sleep (yes/no), and 9 item index measures of sleep disturbance provide composite scores: sleep problem summary, overall sleep problem. Except adequacy, optimal sleep and quantity, higher scores=more impairment. Scores transformed (actual raw score [RS] minus lowest possible score divided by possible RS range*100); total score range:0-100; higher score=more intensity of attribute.
Time Frame: Baseline, Week 21
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 238 | 240
Units on a scale
  Baseline: Sleep Disturbance (n=238, 240) | 29.68 (1.70) | 26.43 (1.70)
  Baseline: Snoring (n=238, 240) | 29.28 (2.31) | 28.09 (2.31)
  Baseline: Awaken Short of Breath (n=238, 240) | 23.64 (2.07) | 19.61 (2.07)
  Baseline: Quantity of Sleep (n=238, 240) | 7.56 (0.11) | 7.59 (0.11)
  Baseline: Adequacy of Sleep (n=238, 240) | 61.30 (2.01) | 63.67 (2.01)
  Baseline: Somnolence (n=238, 240) | 32.29 (1.56) | 29.31 (1.56)
  Baseline: Sleep Problem Index (9) (n=238, 240) | 31.60 (1.32) | 28.15 (1.32)
  Week 21: Sleep Disturbance (n=212, 210) | 24.99 (1.37) | 25.31 (1.39)
  Week 21: Snoring (n=212, 210) | 28.07 (1.89) | 26.12 (1.90)
  Week 21: Awaken Short of Breath (n=212, 210) | 16.26 (1.73) | 18.20 (1.74)
  Week 21: Quantity of Sleep (n=212, 210) | 8.79 (0.17) | 8.77 (0.17)
  Week 21: Adequacy of Sleep (n=212, 210) | 63.87 (1.68) | 64.53 (1.69)
  Week 21: Somnolence (n=212, 210) | 32.04 (1.36) | 29.98 (1.37)
  Week 21: Sleep Problem Index (9) (n=212, 210) | 27.88 (1.04) | 27.54 (1.05)
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Baseline Sleep disturbance: ANCOVA model was used to calculate least square (LS) mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.1160, ANCOVA; LS Mean Difference (Final Values) = 3.25, 95% CI 2-sided [-0.81 to 7.31], Standard Error of Mean 2.07
Statistical Analysis 2: Comparison: Pregabalin vs Gabapentin; Week 21 Sleep disturbance: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.8490, ANCOVA; LS Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-3.62 to 2.98], Standard Error of Mean 1.68
Statistical Analysis 3: Comparison: Pregabalin vs Gabapentin; Baseline snoring: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.6728, ANCOVA; LS Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-4.34 to 6.73], Standard Error of Mean 2.82
Statistical Analysis 4: Comparison: Pregabalin vs Gabapentin; Week 21 snoring: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.3954, ANCOVA; LS Mean Difference (Final Values) = 1.96, 95% CI 2-sided [-2.56 to 6.47], Standard Error of Mean 2.30
Statistical Analysis 5: Comparison: Pregabalin vs Gabapentin; Baseline Awaken Short of Breath: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.1106, ANCOVA; LS Mean Difference (Final Values) = 4.03, 95% CI 2-sided [-0.92 to 8.98], Standard Error of Mean 2.52
Statistical Analysis 6: Comparison: Pregabalin vs Gabapentin; Week 21 Awaken Short of Breath: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.3603, ANCOVA; LS Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-6.09 to 2.22], Standard Error of Mean 2.11
Statistical Analysis 7: Comparison: Pregabalin vs Gabapentin; Baseline Quantity of Sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.8312, ANCOVA; LS Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.30 to 0.24], Standard Error of Mean 0.14
Statistical Analysis 8: Comparison: Pregabalin vs Gabapentin; Week 21 Quantity of Sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.9101, ANCOVA; LS Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.38 to 0.42], Standard Error of Mean 0.20
Statistical Analysis 9: Comparison: Pregabalin vs Gabapentin; Baseline Adequacy of Sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.3346, ANCOVA; LS Mean Difference (Final Values) = -2.37, 95% CI 2-sided [-7.19 to 2.45], Standard Error of Mean 2.45
Statistical Analysis 10: Comparison: Pregabalin vs Gabapentin; Week 21 Adequacy of Sleep: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.7491, ANCOVA; LS Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-4.69 to 3.37], Standard Error of Mean 2.05
Statistical Analysis 11: Comparison: Pregabalin vs Gabapentin; Baseline Somnolence: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.1162, ANCOVA; LS Mean Difference (Final Values) = 2.98, 95% CI 2-sided [-0.74 to 6.71], Standard Error of Mean 1.90
Statistical Analysis 12: Comparison: Pregabalin vs Gabapentin; Week 21 Somnolence: ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.2163, ANCOVA; LS Mean Difference (Final Values) = 2.06, 95% CI 2-sided [-1.21 to 5.32], Standard Error of Mean 1.66
Statistical Analysis 13: Comparison: Pregabalin vs Gabapentin; Baseline Sleep Problem Index (9): ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.0321, ANCOVA; LS Mean Difference (Final Values) = 3.45, 95% CI 2-sided [0.30 to 6.61], Standard Error of Mean 1.61
Statistical Analysis 14: Comparison: Pregabalin vs Gabapentin; Week 21 Sleep Problem Index (9): ANCOVA model was used to calculate LS mean estimates of the treatment difference along with 95% CI, with main effects of treatment and country; for post-baseline, baseline was included as a covariate; Test type: Superiority or Other; p = 0.7889, ANCOVA; LS Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-2.17 to 2.85], Standard Error of Mean 1.28

9. Secondary Outcome: Percentage of Participants With Optimal Sleep Assessed Using Medical Outcomes Study-Sleep Scale (MOS-SS) Score.
Description: MOS-SS: participant-rated 12 item questionnaire to assess constructs of sleep over past week. It included 7 subscales: sleep disturbance, snoring, awakened short of breath, sleep adequacy, somnolence, sleep quantity and optimal sleep. Participants responded whether their sleep was optimal or not by choosing yes or no. Percentage of participants with optimal sleep are reported.
Time Frame: Baseline, Week 21
Population: FAS included all randomized participants who had received at least 1 blinded dose of study drug and had at least 1 baseline and post baseline primary efficacy evaluation. N (number of participants analyzed)=participants who were evaluable for this measure. n=number of participants evaluable at specifictime points for each arm group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Gabapentin
Number analyzed (Participants) | 238 | 240
percentage of participants
  Baseline (n=238, 240) | 49.2 | 58.8
  Week 21 (n=212, 210) | 51.4 | 58.6
Statistical Analysis 1: Comparison: Pregabalin vs Gabapentin; Baseline: Logistic regression model was used to estimate odds ratio and corresponding 95% CI of treatment difference, with treatment as fixed effect and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.0252, Regression, Logistic; Odds Ratio (OR) = 0.653, 95% CI 2-sided [0.449 to 0.948]
Statistical Analysis 2: Comparison: Pregabalin vs Gabapentin; Week 21: Logistic regression model was used to estimate odds ratio and corresponding 95% CI of treatment difference, with treatment as fixed effect and for post-baseline assessments baseline was included as a covariate; Test type: Superiority or Other; p = 0.3459, Regression, Logistic; Odds Ratio (OR) = 0.811, 95% CI 2-sided [0.524 to 1.254]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Gabapentin
Serious Adverse Events (participants affected / at risk) | 13/241 | 14/241
Other Adverse Events (participants affected / at risk) | 77/241 | 77/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=241) | Gabapentin (N=241)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 3 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2
Grand mal convulsion (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Withdrawal syndrome (Psychiatric disorders) | 1 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=241) | Gabapentin (N=241)
Dry mouth (Gastrointestinal disorders) | 12 | 8
Weight increased (Investigations) | 23 | 15
Dizziness (Nervous system disorders) | 22 | 21
Headache (Nervous system disorders) | 21 | 25
Somnolence (Nervous system disorders) | 35 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.